CLINICAL TRIAL: NCT04567303
Title: A Three-part, Phase I/II Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Zifibancimig Following Intravitreal Administration of Multiple Ascending Doses and Continuous Delivery From the Port Delivery in Patients With Neovascular Age-related Macular Degeneration
Brief Title: Study of Zifibancimig in Participants With Neovascular Age-related Macular Degeneration
Acronym: BURGUNDY
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BP41670
Record Dates: First submitted 2020-09-24; First posted 2020-09-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Intervention Model Description: Part 1 of the study will be an open-label multiple ascending dose (MAD) study, followed by subsequent assignment to 2 groups in Part 2. Part 3 will enroll new participants to compare the efficacy of zifibancimig PD implant versus ranibizumab released via the PD implant.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part 1: Visual Acuity (VA) examiner; Part 2: Participant, Investigator, VA examiner and Sponsor; Part 3: Participant, Investigator, VA examiner and Sponsor.
  The sponsor and its agents have been unblinded to treatment assignment in Parts 2 and 3, as of protocol amendment version 12.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (6):
- Part 1: IVT Injections (Experimental): Zifibancimig administered in multiple ascending dose levels through IVT injections.
  Interventions: Drug: Zifibancimig
- Part 2: PD With High Dose (Experimental): Zifibancimig administered at a high dose through the PD implant, followed by ranibizumab, 100 milligrams per milliliter (mg/mL), administered through the PD implant.
  Interventions: Drug: Zifibancimig; Drug: Ranibizumab; Device: Port Delivery Platform
- Part 2: PD With Low Dose (Experimental): Zifibancimig administered at a low dose through the PD implant, followed by ranibizumab, 100 mg/mL, administered through the PD implant.
  Interventions: Drug: Zifibancimig; Drug: Ranibizumab; Device: Port Delivery Platform
- Part 3: PD With High Dose (Experimental): Zifibancimig administered at a high dose through the PD implant, followed by ranibizumab, 100 mg/mL, administered through PD implant.
  Interventions: Drug: Zifibancimig; Drug: Ranibizumab; Device: Port Delivery Platform
- Part 3: PD With Low Dose (Experimental): Zifibancimig administered at a low dose through the PD implant, followed by ranibizumab, 100 mg/mL, administered through PD implant.
  Interventions: Drug: Zifibancimig; Drug: Ranibizumab; Device: Port Delivery Platform
- Part 3: PD With Ranibizumab (Active Comparator): 100 mg/mL of ranibizumab administered through the PD implant.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Zifibancimig — Part 1: multiple ascending doses by IVT injection. Each participant will receive zifibancimig at a constant volume of 50 microliter (µL) in the study eye.
  Part 2: participants will be randomized to one of two dose levels of zifibancimig in the PD implant.
  Part 3: Participants will receive one of the two dose levels of zifibancimig in the PD implant.
  Other Names: RO7250284
  Arms: Part 1: IVT Injections; Part 2: PD With High Dose; Part 2: PD With Low Dose; Part 3: PD With High Dose; Part 3: PD With Low Dose
Drug: Ranibizumab — Participants will receive ranibizumab 100 mg/mL through the PD implant
  Arms: Part 2: PD With High Dose; Part 2: PD With Low Dose; Part 3: PD With High Dose; Part 3: PD With Low Dose; Part 3: PD With Ranibizumab
Device: Port Delivery Platform — Participants will receive intraocular refillable device that is surgically inserted into the eye for continuous delivery of drugs into the vitreous.
  Arms: Part 2: PD With High Dose; Part 2: PD With Low Dose; Part 3: PD With High Dose; Part 3: PD With Low Dose

SUMMARY:
This is a first in-human study to investigate the safety, tolerability and efficacy of zifibancimig administered through intravitreal (IVT) injections and via the port delivery (PD) implant in participants with neovascular age-related macular degeneration (nAMD).

ELIGIBILITY:
Part 1, Part 2 and Part 3

Inclusion Criteria:

* Willing to allow AH collection

Part 1 and Part 2

Ocular Inclusion Criteria for Study Eye:

* Choroidal neovascularization (CNV) exclusively due to age-related macular degeneration (AMD)
* Anti-vascular endothelial growth factor (VEGF) or anti-VEGF/Angiopoietin-2 (Ang-2) IVT treatment-naïve, or pre-treated with anti-VEGF or anti-VEGF/Ang-2 no less than two months prior to Day 1
* Sufficiently clear ocular media and adequate pupillary dilatation to allow for analysis and grading by the central reading center of fundus photography (FP), fluorescein angiography (FA), fundus autofluorescence (FAF), and spectral domain optical coherence tomography (SD-OCT) images
* Decreased BCVA attributable primarily to nAMD, with BCVA letter score of 78 to 34 letters (inclusive) on ETDRS-like charts at screening. In case both eyes of a participant are eligible, the eye with the lower BCVA score should become the study eye

Part 3

Ocular Inclusion Criteria for Study Eye:

* CNV exclusively due to AMD
* Diagnosis of nAMD within 36 months prior to the screening visit
* Previous treatment with at least one IVT anti-VEGF or anti-VEGF/Ang-2 administrations IVT for nAMD. The last IVT administration must have occurred at least 21 days prior to the screening visit
* Demonstrated response to prior IVT anti-VEGF or anti-VEGF/Ang-2 treatment since diagnosis
* Availability of historical VA data prior to the first anti-VEGF or anti-VEGF/Ang-2 treatment for nAMD
* Sufficiently clear ocular media and adequate pupillary dilatation to allow for analysis and grading
* Decreased BCVA attributable primarily to nAMD with letter score of 78 to 34 letters (inclusive) or better on ETDRS-like charts

Ocular Exclusion Criteria for Study Eye:

* History of vitrectomy surgery, submacular surgery, other intraocular surgery, or any planned surgical intervention during the study period
* Cataract surgery without complications within three months preceding the screening visit or planned during the study period
* Aphakia or absence of the posterior capsule. Previous violation of the posterior capsule is also an exclusion criterion, unless it occurred as a result of yttrium-aluminum garnet laser posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation
* Prior macular treatment with verteporfin, external beam radiation therapy, transpupillary thermotherapy, or any type of laser photocoagulation
* Prior treatment with IVT corticosteroids or implant (e.g., triamcinolone, ozurdex, iluvien)
* Subretinal hemorrhage >50% of the total lesion area and/or involving the fovea
* Subfoveal fibrosis or subfoveal atrophy
* Retinal pigment epithelial tear involving the macula
* History of vitreous hemorrhage, rhegmatogenous retinal detachment, glaucoma-filtering surgery, tube shunts, or microinvasive glaucoma surgery, and corneal transplant
* History of rhegmatogenous retinal tears or peripheral retinal breaks within three months prior to the screening visit
* Actual or history of myopia >-8 diopters
* Uncontrolled ocular hypertension or glaucoma (defined as intraocular pressure [IOP] >25 millimeters of mercury (mm Hg) or a cup to disc ratio >0.8, despite treatment with antiglaucoma medication) and any such condition the Investigator determines may require a glaucoma-filtering surgery during a participant's participation in the study
* Concurrent intraocular conditions (e.g., cataract, diabetic retinopathy, epiretinal membrane with traction, macular hole) that, in the opinion of the Investigator, could either: require medical or surgical intervention during the study period to prevent or treat visual loss that might result from that condition; or likely contribute to loss of BCVA over the study period if allowed to progress untreated; or preclude any visual improvement due to substantial structural damage
* Concurrent conjunctival, Tenon's capsule, and/or scleral condition in the supero-temporal quadrant of the eye (e.g., scarring, thinning, mass) that may affect the implantation, subsequent tissue coverage, and refill-exchange procedure of the PD implant
* Prior treatment with any medication for geographic atrophy (GA) during the last 3 months prior to screening
* Prior treatment with any anti-VEGF-C or anti-VEGF-D inhibitors

Exclusion Criteria for Fellow Eye

* BCVA letter score using ETDRS charts of < 34 letters
* Treatment with IVT anti-VEGF or anti-VEGF/Ang-2 agents within one week prior to Day 1 (concurrent treatment with SUSVIMO^TM in the fellow eye is not exclusionary)

Exclusion Criteria for Either Eye

* CNV due to causes other than nAMD, such as ocular histoplasmosis, trauma, pathological myopia, angioid streaks, choroidal rupture, uveitis or central serous chorioretinopathy
* Prior participation in a clinical trial involving anti-VEGF drugs within six months prior to the screening visit, other than ranibizumab, aflibercept, or faricimab including approved biosimilars
* Active intraocular inflammation (grade trace or above), infectious conjunctivitis, keratitis, scleritis, or endophthalmitis
* History of uveitis, including history of any intraocular inflammation following intravitreal therapy
* Prior treatment with brolucizumab
* Prior gene therapy for nAMD

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Ocular and Systemic (Non-ocular) Adverse Events (AEs) | Part 1: Baseline up to Week 24; Parts 2 & 3: Baseline up to Week 48
Percentage of Participants With Ocular AEs During the Post-operative and Follow-up Periods | Parts 2 and 3: From Day 1 to Week 4 and during follow-up period (up to Week 48)
Percentage of Participants With Adverse Events of Special Interest (AESIs) Including Ocular AESIs | Part 1: Baseline up to Week 24; Parts 2 and 3: Baseline up to Week 48
Percentage of Participants With Ocular AESIs During the Post-operative and Follow-up Periods | Parts 2 and 3: From Day 1 to Week 4 and during follow-up period (up to Week 48)
Duration of Ocular AESIs | Part 1: Baseline up to Week 24; Parts 2 and 3: Baseline up to Week 48
Duration of Ocular AESIs During the Post-operative and Follow-up Periods | Parts 2 and 3: From Day 1 to Week 4 and during follow-up period (up to Week 48)
Percentage of Participants With Adverse Device Effects (ADEs) | Parts 2 and 3: Baseline up to Week 48
Duration of ADEs | Parts 2 and 3: Baseline up to Week 48
Percentage of Participants With Anticipated Serious ADEs (ASADEs) | Parts 2 and 3: Baseline up to Week 48
Duration of ASADEs | Parts 2 and 3: Baseline up to Week 48
Change From Baseline in Early Treatment Diabetic Retinopathy Study - Best Corrected Visual Acuity (ETDRS-BCVA) Score at Week 48 | Part 3: Baseline (baseline visit, before implant insertion), and Week 48
  ETDRS-BCVA will be used to quantify visual acuity. BCVA is measured using an eye chart and is reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Zifibancimig in Blood and Aqueous Humor (AH) | Part 1: Baseline up to Week 24; Parts 2 and 3: Baseline up to Week 144
Time of Maximum Concentration Observed (Tmax) of Zifibancimig in Blood and AH | Part 1: Baseline up to Week 24; Parts 2 and 3: Baseline up to Week 144
Concentration at the End of a Dosing Interval Before the Next Dose Administration (Ctrough) of Zifibancimig in Blood and AH | Part 1: Baseline up to Week 24; Parts 2 and 3: Baseline up to Week 144
Area Under the Curve (AUC) of Zifibancimig in Blood and AH | Part 1: Baseline up to Week 24; Parts 2 and 3: Baseline up to Week 144
Percentage of Participants Who did not Meet Supplemental Treatment Criteria for the PD Implant With Zifibancimig | Part 3: Week 36, Week 40, and Week 44
Percentage of Participants Who Gained or Lost ≥15, ≥10 ≥5 or ≥0 Letters in ETDRS-BCVA Score From Baseline to Week 48 | Part 3: Baseline to Week 48
  ETDRS-BCVA will be used to quantify visual acuity. BCVA is measured using an eye chart and is reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Change From Baseline in Central Subfield Thickness (CST) at Week 48 | Part 3: Baseline, and Week 48
Change From Baseline Over Time in CST | Part 3: Baseline to end of follow-up period (up to Week 144)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (48):
- United States (47):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - The Retina Partners, Encino, California
  - Retinal Consultants Med Group, Sacramento, California
  - Orange County Retina Med Group, Santa Ana, California
  - Macula Retina Vitreous Research Institute, Torrance, California
  - Southwest Retina Consultants, Durango, Colorado
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Maine Eye Center, Portland, Maine
  - The Retina Care Center, Baltimore, Maryland
  - Johns Hopkins Med, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Associated Retinal Consultants, Royal Oak, Michigan
  - VitreoRetinal Surgery, PLLC., Saint Louis Park, Minnesota
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - NJ Retina - Teaneck, Teaneck, New Jersey
  - Retina Vit Surgeons/Central NY, Liverpool, New York
  - Long Is. Vitreoretinal Consult, Westbury, New York
  - Duke Eye Center, Durham, North Carolina
  - Graystone Eye, Hickory, North Carolina
  - OSU Eye Physicians & Surgeons, Columbus, Ohio
  - Mid Atlantic Retina - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Charleston Neuroscience Inst, Ladson, South Carolina
  - Carolina Eyecare Physicians, Mt. Pleasant, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Southeastern Retina Associates, Knoxville, Tennessee
  - Tennessee Retina PC., Nashville, Tennessee
  - Austin Research Center for Retina, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Texas, Houston, Texas
  - Brown Retina Institute, San Antonio, Texas
  - Retina Center of Texas, Southlake, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Kapoor Institute, Norfolk, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington
- Emanuelli Research and Development Center LLC, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing